CLINICAL TRIAL: NCT05996835
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Four-arm, Parallel-group, Dose-finding Phase 2b Study to Investigate the Safety and Efficacy of TIN816 Via a Single Intravenous Infusion in the Treatment of Participants With Sepsis-associated Acute Kidney Injury (CLEAR-AKI)
Brief Title: Phase 2b Study to Investigate the Safety and Efficacy of TIN816 in Sepsis-associated Acute Kidney Injury (CLEAR-AKI)
Acronym: CLEAR-AKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTIN816B12202
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury Due to Sepsis
Keywords: Sepsis; acute kidney injury; anti-inflammatory; immunosuppression; intensive care unit
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TIN816 Dose A (Experimental): Administered as a one time intravenous dose
  Interventions: Biological: TIN816 70 mg lyophilisate powder
- TIN816 Dose B (Experimental): Administered as a one time intravenous dose
  Interventions: Biological: TIN816 70 mg lyophilisate powder
- TIN816 Dose C (Experimental): Administered as a one time intravenous dose
  Interventions: Biological: TIN816 70 mg lyophilisate powder
- Placebo (Placebo Comparator): 0.9% sterile saline administered as a one time intravenous dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TIN816 70 mg lyophilisate powder — Immunotherapy Recombinant human CD39 enzyme
  Arms: TIN816 Dose A; TIN816 Dose B; TIN816 Dose C
Other: Placebo — 0.9% sterile saline solution
  Arms: Placebo

SUMMARY:
The purpose of this Ph2b study is to characterize the dose-response relationship and to evaluate the safety and efficacy of three different single doses of TIN816 in hospitalized adult participants in an intensive care setting with a diagnosis of sepsis-associated acute kidney injury (SA-AKI).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, four-arm, parallel-group, dose-finding phase 2b study. The study will enroll hospitalized adult participants with a diagnosis of sepsis and acute kidney injury (AKI). The study consists of a screening period (24-48 hours), a treatment period (Day 1), and post-treatment period (Day 2 to 90). Screening will take place during hospitalization in ICU (or intermediate care unit/HDU) where potential participants will undergo screening to assess the presence of sepsis and AKI. At Treatment Day 1, participants who meet eligibility criteria at screening and baseline will be randomized in a 3:1:1:3 ratio to receive a one-time treatment of TIN816 or placebo by intravenous infusion in a participant and investigator-blinded fashion. Treatment Day 1 is followed by a 90-day post-treatment period for safety and efficacy assessments. An interim analysis (IA) is planned when approximately 120 participants complete Day 30 visit. A final analysis will be performed after all participants have completed Day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained in accordance with local regulations.
2. ≥ 18 to ≤ 85 years of age
3. Admitted to ICU or intermediate care unit/ high dependency care unit (HDU)
4. Diagnosis of sepsis according to criteria defined by The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) based on:

   * Suspected or confirmed infection AND
   * Acute increase of SOFA score of 2 or more (excluding renal component). The baseline SOFA score should be assumed to be zero unless the participant is known to have pre-existing (acute or chronic) organ dysfunction before the onset of infection
5. Diagnosis of AKI Stage 1 or greater per the following criterion at randomization:

An absolute increase in serum or plasma creatinine by ≥ 0.3 mg/dL (≥ 26.5 µmol/L) within 48 hours or presumed to have occurred in the previous 48 hours as compared to the reference serum creatinine.

* For participants with hospital-acquired AKI, a stable serum creatinine obtained in the hospital prior to AKI diagnosis should be used as the reference serum creatinine.
* For participants presenting from community, the reference serum creatinine should be estimated using the following order of preference:

  1. The most recent value within 3 months of the hospital admission. If not available:
  2. The most recent value between 3 and 12 months prior to hospital admission. If not available:
  3. At hospital admission

Exclusion criteria

1. Not expected to survive for 24 hours
2. Not expected to survive for 30 days due to medical conditions other than SA-AKI
3. History of CKD with a documented estimated GFR <30 mL/min prior to admission to hospital
4. eGFR <45mL/min at admission without any other reference serum eGFR within last 12-months
5. Receiving RRT or a decision has been made to initiate RRT within 24 hours after randomization
6. Weight is less than 40 kg or more than 125 kg.
7. Limitations to the use of mechanical ventilation, RRT or vasopressors/inotropes (N.B. limitations on Cardiopulmonary resuscitation (CPR)e.g., do-not-resuscitate orders are not an exclusion criterion unless associated with likely poor outcome in next 24 hours)
8. Sepsis diagnosis according to sepsis inclusion criteria for a period longer than 72 hours prior to ICU admission
9. AKI diagnosis according to AKI inclusion criteria over 48 hours after admission to ICU
10. Inability to administer study drug within 24 hours of diagnosis of AKI according to AKI inclusion criteria
11. Presence of AKI, in the Investigator's opinion, as suggested by clinical manifestation, e.g., prolonged oliguria or severe renal dysfunction on admission without a history of CKD, for a period longer than 24 hours prior to study drug administration
12. Evidence of recovery from AKI based on the investigator's clinical judgement prior to randomization
13. AKI is most likely attributable to other causes than sepsis, such as nephrotoxic drugs (Non-steroidal anti-inflammatory drugs (NSAIDs), contrast, aminoglycosides, etc.) or renal perfusion-related (acute abdominal aortic aneurysm, dissection, renal artery stenosis), urinary obstruction
14. Documented (biopsy proven) or suspected history of acute or sub-acute kidney diseases such as rapidly progressive glomerular nephritis (RPGN) and acute interstitial nephritis (AIN)
15. Patients who are post-nephrectomy
16. Patients with permanent incapacitation
17. Patients who are thrombocytopenic at screening (platelet count <50,000 per microliter) who have active/uncontrolled bleeding or who present current or past conditions indicating high risk for bleeding in the opinion of the investigator (e.g. coagulopathies, previous history of major non-traumatic bleeding etc.)
18. Immunosuppressed patients

    * History of immunodeficiency diseases
    * Receiving immunosuppressant treatment or on chronic high doses (high-dose therapy exceeding 2 weeks of treatment) of steroids equivalent to prednisone/prednisolone 0.5 mg/kg/day, including solid organ transplant patients. Patients with septic shock treated with corticosteroids (as per the Surviving Sepsis Guidelines) can be included.
19. Patients with known or presumed latent or active TB based on clinical history or imaging e.g. patients on TB preventive therapy or close/household contacts of pulmonary TB patients
20. Known active hepatitis B or C infection (clinical diagnosis or positive infection serology), or advanced chronic liver disease, confirmed by a Child-Pugh score of 10-15 (Class C)
21. Acute pancreatitis with no established source of infection
22. Active hematological malignancy (previous hematological malignancies that are not actively treated are allowable)
23. Burns requiring ICU treatment
24. Sepsis attributed to confirmed COVID-19
25. Use of other investigational drugs within 5 half-lives of enrollment, within 30 days (e.g., small molecules) or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations
26. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes
27. Any medical conditions that could significantly increase risk of participants' safety by participating in this study according to investigator's judgement
28. Women with a positive pregnancy test, pregnancy or breast feeding
29. Women of childbearing potential, unless they are using highly effective methods of contraception for the entire duration of the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Average of area under the time-corrected creatinine clearance curve (AUC1-8) | Day 1 to Day 8
  The weighted average of area under the time-corrected endogenous creatinine clearance curve.
  Urine volume, urinary creatinine, and the serum creatinine measurements will be used for calculation. Day 1-8 measurements will be included.

SECONDARY OUTCOMES:
Percentage of participants with major adverse kidney events (MAKE) | Day 1 to Day 90
  A binary composite endpoint of major adverse kidney events (MAKE) including death, use of Renal Replacement Therapy (RRT) and ≥25% reduction from reference in estimated Glomular Filtration Rate (eGFR) at Day 90.
Area under the time-corrected endogenous serum creatinine curve for Day 1 to Day 14 and Day 1 to Day 30. | Day 1 to Day 14 and Day 1 to Day 30
  The weighted average of area under the time-corrected endogenous serum creatinine curve from Day 1 to Day 14 and Day 1 to Day 30.
Area under the time-corrected endogenous serum cystatin C curve for Day 1 to Day 14 and Day 1 to Day 30 | Day 1 to Day 14 and Day 1 to Day 30
  The weighted average of area under the time-corrected endogenous serum cystatin-C curve from Day 1 to Day 14 and Day 1 to Day 30.
Area under the time-corrected creatinine clearance curve (AUC5-14) | Day 5 to Day 14
  The weighted average of area under the time-corrected endogenous creatinine clearance curve.
  Urine volume, urinary creatinine, and the serum creatinine measurements will be used for calculation. Day 5-14 measurements will be included.
Percentage of participants who had renal replacement therapy (RRT) from Day 1 to Day 90 | Day 1 to Day 90
  Use of RRT at any time during the treatment period will be reported.
Percentage of participants with RRT dependency at Day 90 | Day 90
  Use of RRT dependency at Day 90 will be reported
Number of days participants alive and free of RRT from Day 1 to Day 90 | Day 1 to Day 90
  Participants who are alive and free of RRT, defined as any participant receiving any form of RRT, will be reported.
Change in Kidney disease improving global outcomes (KDIGO) score from Baseline to Day 14 | 14 Days
  The KDIGO classification system stages AKI into three levels based on serum creatinine elevation in parallel with degree and duration of oliguria. Participants are classified based on the worst finding (either serum creatinine or oliguria). The stages range from 1-3, with higher scores indicating the most severe stage of AKI.
Percentage of participants with ≥25% reduction in eGFR at Day 90 | 90 Days
  Percentage of participants with ≥ 25% reduction from reference to Day 90.
Mean change of sequential organ failure assessment score (SOFA) from baseline to Day 30 | 30 Days
  The SOFA score was developed to assess the acute morbidity of critical illness at a population level. The score is routinely calculated on admission to ICU and at each 24-hour period that follows. It is composed of six criteria which reflect the function of a specific organ system (respiratory, cardiovascular, renal, neurological, hepatic and hematological) and allocates a score of 0-4.
  Scores ranges from 0-24, with higher scores indicating greater dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (114):
- United States (24):
  - University Of Alabama, Birmingham, Alabama
  - UC San Francisco Medical Center, San Francisco, California
  - Stanford Healthcare, Stanford, California
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Northwestern Memorial Hospital, Evanston, Illinois
  - Endeavor Health, Glenview, Illinois
  - Univ Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Good Samaritan Hospital, Corvallis, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - U Of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Baylor Scott and White, Dallas, Texas
  - Utah Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Providence Med Resch Center and Chindren Hosp, Spokane, Washington
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Pilar, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Santa Fe
- Australia (2):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Heidelberg, Victoria
- Novartis Investigative Site, Innsbruck, Tyrol, Austria
- Belgium (4):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Ottignies
- Brazil (5):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (6):
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Wuhan
- France (11):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Garches
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster
- Hungary (4):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Székesfehérvár
- India (5):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
- Italy (7):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (12):
  - Novartis Investigative Site, Kamogawa, Chiba
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ureshino, Saga-ken
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kumamoto
- Novartis Investigative Site, Pretoria, South Africa
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
- United Kingdom (4):
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com